CLINICAL TRIAL: NCT03756831
Title: The Influence of BMI on Core Stability in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wafaa Mahmoud Amin (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Wafaa Mahmoud Amin, Principal Investigator, University of Jazan
Organization: University of Jazan (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2378388561
Record Dates: First submitted 2018-11-23; First posted 2018-11-28 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Overweight and Obesity; Balance; Distorted
Keywords: BMI, Core Stability, Healthy Adult
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: 3x3 factorial design, according to body mass index (Independent variable)subjects will be divided into three groups (Group I - normal subjects-BMI<25 kg/m2, Group II -overweight subjects-BMI, 25-30 kg/m2), Group III -obese subjects- BMI>30 kg/m2). Core stability (dependent variable) will be measured by three tests : bilateral static balance with open and close eye, uni-pedal static balance test, and dynamic balance test using Prokin System for balance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (normal subjects) (Active Comparator): 30 individuals (15 male, and 15 female students) with (BMI<25 kg//m^2)). Core Stability Assessment will be performed for them using Prokin system.
  Interventions: Diagnostic Test: Core Stability Assessment
- Group II (overweight subjects) (Active Comparator): 30 individuals (15 male, and 15 female students) with (BMI, 25-30 kg//m^2)). Core Stability Assessment will be performed for them using Prokin system.
  Interventions: Diagnostic Test: Core Stability Assessment
- Group III (obese subjects) (Active Comparator): 30 individuals (15 male, and 15 female students) (BMI>30 kg//m^2)). Core Stability Assessment will be performed for them using Prokin system.
  Interventions: Diagnostic Test: Core Stability Assessment

INTERVENTIONS:
Diagnostic Test: Core Stability Assessment — Core Stability Assessment will be consisted of bilateral static balance with open and close eye, right foot balance test, and dynamic balance test.
  Other Names: Balance Assessment

SUMMARY:
This study will be conducted to investigate the influence of body mass index (BMI) on core stability (CS) in healthy subjects. The participants in this study will be 90 healthy subjects with right dominant lower limb (49 females and 49 males) they will be recruited from College of Applied Medical Sciences, Jazan University.

DETAILED DESCRIPTION:
Subjects will be categorized according to BMI into three groups:

Group I (normal subjects): 30 individuals (15 male, and 15 female students) with (BMI<25 kg//m^2)) Group II (overweight subjects): 30 individuals (15 male, and 15 female students) with (BMI, 25-30 kg//m^2)).

Group III (obese subjects): 30 individuals (15 male, and 15 female students) (BMI>30 kg//m^2)).

Motor control element of CS will be investigated by assessing bilateral static balance with open and close eye, right foot balance test, and dynamic balance test using Prokin System for balance. Data of this study will be statistically analyzed by performing descriptive (Mean and standard deviation) and inferential statistics (One way ANOVA, Unpaired T test) at level of significance p=<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects would not have any diseases of the central nervous system.
2. Subjects would not have any orthopedic disorders either of the trunk or the lower limbs in the previous year.
3. None of the subjects has history of balance training ( Erkmen et al., 2010, Li Li, 2012) .

Exclusion Criteria:

1. Sign of foot pain, reduced tactile and thermal foot sensibility.
2. Peripheral neuropathy.
3. A history of previous back or abdominal surgery/injury
4. A history of patellofemoral pain syndrome, plantar fasciitis, and back pain .
5. Limb-length discrepancy, and anterior or posterior tibialis dysfunction.
6. Evidence of a systemic or musculoskeletal disease within the past six months (AlAbdulwahab & Kachanathu, 2016).

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Static balance test with eyes opened | 30 Seconds
  After explaining the tests to the subjects, data will be entered and the device will be calibrated. Both feet of the subjects will be placed on the balance platform nakedly with eyes are opened.
Static balance test with eyes closed | 30 Seconds
  After explaining the tests to the subjects, data will be entered and the device will be calibrated. Both feet of the subjects will be placed on the balance platform nakedly with eyes closed.
Unipedal static balance | 30 Seconds
  It will be measured respectively on right foot with eyes are opened.
Dynamic (Equilibrium/ Disequilibrium test) | 60 Seconds
  the subject will stand on right foot(dominant), and see some galleries that come against. The subject's scope is to enter into those galleries and to maintain the tilting board as firm as possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Riyadh, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided